CLINICAL TRIAL: NCT04713995
Title: The Role of the Gut Microbiome in Axial Spondyloarthritis (AxSpA) Disease Activity
Brief Title: Microbiome and Axial Spondyloarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sufficient samples and data have been collected for data analyses.
Sponsor: Viome (Industry)
Collaborators: Spondylitis Association of America (SAA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: V150
Record Dates: First submitted 2020-08-31; First posted 2021-01-19 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Axial Spondyloarthritis
Keywords: AxSpA; Microbiome; Viome; ASDAS; AS; Spondyloarthritis; HbA1c; Ankylosing; HLA B27; Spine; Ankylosing Spondylitis
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylarthritis; Spondylitis, Ankylosing

STUDY DESIGN:
Intervention Model Description: 400 Participants are enrolled and paired matching for HLA-B27+ and control (mASDAS <1.3) and case group (mASDAS = or > 1.3) and compared to a healthy control group. Samples and surveys are collected from all participants. Then again at 3 months and 6 months if they agree to complete the longitudinal arms of the study.
Masking Description: All recruitment happens online. All nutritional recommendations look the same, but may be different between participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Study Participants (Other): Enrolled with: AxSpA diagnosis, HLA-B27 positive, mASDAS > or = 1.3 and HLA-B27 positive. Will complete surveys online or on an app, about mental and physical health and how they are doing, submits and collection of samples (blood, stool, saliva, urine, fasting blood test at local lab). Receives results of some of the analysis of samples. Participants that qualify and complete the first set of samples can be eligible for the 3 and 6 month longitudinal follow-up collection kits.
  All participants receive dietary recommendations based on samples collected and the analysis of the microbiome.
  Interventions: Other: Dietary recommendations

INTERVENTIONS:
Other: Dietary recommendations — Dietary recommendations based on microbiome analysis of samples will be given and expected to receive and report in ~3 months survey after following recommendations.

SUMMARY:
The purpose of this interventional study is to identify the root cause(s) of AxSpA (Axial Spondyloarthritis) relapses, which are likely due to the combination of nutrition, gut microbiome activities, leaky gut, and human genes (particularly from the immune system). This will be done by identifying molecular features of the microbiome that are associated with AxSpA flares, progression and relapses.

The study will recruit participants with confirmed AxSpA diagnosis and who are HLA-B27 positive. During screening potential participants allow access to medical records to confirm eligibility requirements, such as diagnosis. Once enrolled, collection kits are sent to participants to collect samples using at-home collection kits and then provide a fasting blood sample at a local lab. Samples are then analyzed to identify features that likely cause AxSpA issues. Survey's are also answered to collect additional health data. Scientists will then use the data to identify the features that likely cause AxSpA flares and relapses.

DETAILED DESCRIPTION:
This is an Interventional study to help find the root causes of AxSpA relapses, flares and progression. The study will enroll 400 participants who are aged 18 or over, are HLA-B27 positive, have had a diagnosis of AxSpA. An informed consent form is acknowledged and medical release signed (to confirm eligibility criteria). Participants sign up online and answer questions about their physical and mental health and how they are doing (through an app and/or website). The participants will be in the study approximately 3 months, unless they agree to complete the 3 and 6 month timeline assessments for the longitudinal timelines, then the study will be completed after those timelines.

If eligible, participants are shipped at-home collection kits which include: saliva, finger-prick blood and stool. A Genova urine test is also included to check intestinal permeability. Participants also make an appointment and go to a local lab to collect an additional blood sample. All samples are shipped via pre-paid mailers. All collections are done within a 1-week window (or 7 days). Clinical samples are collected in order to analyze specific molecular features associated with AxSpA in the microbiome found in participants.

After shipping home collection kits and visiting the lab for a blood draw, participants receive diet recommendations which they will follow for ~3 months, after which time they will fill out a study survey to complete the first timeline in the study.

If interested in participating in the longitudinal portion of the study, participants can also complete the 3-month and 6-month home collection, blood collection at the local lab and additional surveys.

Scientists hope to find the microbiome and molecular information that corresponds to flares, health and wellness in the microbiome in patients with AxSpA.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 disease code or diagnosis for AxSpA
* Confirmed diagnosis of AxSpA, based on ASDAS criteria including both non-radiographic axial spondyloarthritis and ankylosing spondylitis
* HLA-B27 positive
* Signed informed consent prior to any study-specific procedures are performed
* Females and males aged 18 years or older
* Able to read, speak and understand English
* Willing and able to use the at-home collection kits and mail in pre-paid mailers
* Willing and able to use a smartphone app or web app to answer surveys
* Willing and able to make and keep/travel to a local lab visit for blood collection
* Willing and able to follow the study instructions, as described in the recruitment letter

Exclusion Criteria:

* Unable or unwilling to use Viome's App on an iPhone or Android smartphone
* Not HLA-B27 positive
* No diagnosis for AxSpA/AS
* Pregnant or nursing
* Other diagnosis of arthritis (rheumatoid, osteoarthritis, psoriatic arthritis, psoriatic spondyloarthritis)
* IBD/Crohn's disease/ulcerative colitis
* Use of antibiotics or Sulfasalazine within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
AxSpA (Axial Spondyloarthritis) disease activity | 1 year
  Analysis using lab results and AI learning models to correspond microbiome activity will be used to see if nutrition affects disease activity of the microbiome of people with AxSpA

CONTACTS AND LOCATIONS:
Overall Officials: Momochilo Vuyisich, PhD, Principal Investigator — Viome Research Institute
Locations (1):
- Viome Research Institute online: https://www.viome.com/VRI/studies, Bothell, Washington, United States

IPD SHARING:
Plan to Share IPD: No